CLINICAL TRIAL: NCT04358757
Title: An Observational Study to Determine Immune and Physical Recovery Following Elective Cesarean Delivery
Brief Title: Immune and Physical Recovery Following Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, PSultan, Associate Professor, Stanford University
Other Study IDs: 51414
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Cesarean Delivery
Keywords: elective cesarean delivery; predictors; recovery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Leucocytes collected will be batch stored and then analysed once al samples collated after study recruitment completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cesarean patients: participants undergoing elective cesarean will have measures of recovery assessed (patient-reported outcome measures and activity data from watch)
  Interventions: Procedure: Elective cesarean delivery

INTERVENTIONS:
Procedure: Elective cesarean delivery — scheduled cesarean delivery for maternal / obstetric indications

SUMMARY:
Pregnancy results in an altered immune state compared to the nonpregnant population. A significant proportion of women undergoing cesarean delivery recover poorly. The first step to determining whether this is an immune driven / associated process is to characterise what effects this surgery has on maternal immune function. "Normal" changes will be evaluated in maternal immune function and activity precipitated by surgery and delivery of the neonate. Immune response to surgery will be compared to historical immune data from patients undergoing non-obstetric surgery (orthopaedic patients).

DETAILED DESCRIPTION:
Variations will be evaluated in baseline and postpartum leukocyte subset distribution and singling pathways within leukocyte subsets (including response to surgery) in women undergoing elective cesarean delivery compare to patients undergoing nonobstetric surgery (orthopaedic data from a completed study). This will help to determine whether baseline immune function and response to trauma (surgery) is the same in the pregnant and non-pregnant states. Women will also be evaluated for clinical recovery parameters using validated scoring measures and objective measurement of physical activity through use of a smartwatch (actigraph) around the peripartum period. This information is of significant importance as it brings us one step closer to identifying immune mechanisms that may be involved in or associated with poorer postpartum recovery.

Aim- to determine whether perioperative immune function can predict women who are likely to have delayed physical recovery or recover poorly as demonstrated by lower scores on subjective clinical questionnaires and collected via watch actigraphy. This will help to determine whether a pre-existing deficient immune state is responsible for a worse recovery profile, which could be identified preoperatively. Similarly whether an impairment in response to surgery is demonstrable, which predisposes women to worse recovery profiles will be evaluated.

Ultimately, earlier identification of at-risk parturients (for example, through a preoperative bedside test) may lead to earlier interventions / patient centred care, in an attempt to improve their recovery trajectory and patient experience.

ELIGIBILITY:
Inclusion Criteria:

* elective cesarean delivery at Lucile Packard Hospital
* age >20 to <50 years old,
* single pregnancy term
* gestational age 37-41 weeks pregnancy,
* elective cesarean delivery,
* spinal or combined spinal-epidural anesthesia as primary anesthesia mode,
* multimodal analgesia regimen (including intrathecal morphine and regular acetaminophen and NSAIDs), single center at Stanford.
* ASA grade 1 or 2.
* gestational diabetes (not requiring insulin or diabetes medications and pre-eclampsia (without severe features) will be included.
* ethnic background: all ethnic backgrounds will be included gender: pregnant women only

Exclusion Criteria:

* refusal to participate

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Elective cesarean delivery
Study Population: women delivering via scheduled cesarean delivery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2023-09-23 (Actual); Study Completion 2023-12-23 (Actual)

PRIMARY OUTCOMES:
Incidence of immune changes from preoperative to day 1 postoperative | immediately prior to surgery versus morning following surgery (approximately 24 hrs apart)
  immune changes include: leukocyte subset distribution, intracellular signaling pathway activity within leukocyte subsets and cytokine-induced responses to ex-vivo stimulation in leukocyte subsets
change in activity (measured by actigraphy) before and after cesarean | 2 weeks pre to 6 weeks postoperative
  Actigraph smartwatch data will be used to assess how activity changes around the time of delivery and determine physical recovery profiles following elective cesarean delivery. Time to baseline and time to plateau of maximal physical activity will be assessed in the postpartum period up to 6 weeks postoperatively.

SECONDARY OUTCOMES:
perioperative response to cytokine stimulation | preoperative, day 1 (and in a subset PACU, umbilical vein, and day 2)
  cytokine stimulation of leucocytes from parturients will be assessed using mass cytometry.
  blood samples will be taken from all participants preoperatively and on morning following surgery.
  10 women will also have: postanesthetic care unit blood, umbilical vein blood and day 2 blood samples taken
ex-vivo leucocyte response | preoperative, day 1 (and in a subset PACU, umbilical vein, and day 2)
  Leucocytes will be chemically stimulated ex-vivo
  for each leukocyte subset, plot stimulated and unstimulated levels and delta (change) in levels at each time point
  10 women will also have: postanesthetic care unit blood, umbilical vein blood and day 2 blood samples taken
immune predictors of delayed physical recovery | preoperative to 6 weeks postoperative
  phenotype (immune profile) associated with delayed physical recovery. determine whether any preoperative immune phenotype (preoperative changes in immune response to chemical stressors) can predict worse activity profiles analysed using actigraph data.
Change in ObsQoR-10 | postoperatively on day 1 and day 2
  relationship between immune markers, actigraphy data using ObsQoR-10 (obstetric quality of recovery -10 item score- validated overall quality of recovery measure)
Change in PROMIS-29 score | postoperatively on week 3 and 6 and 3 months
  relationship between immune markers, actigraphy data using PROMIS-29 (validated overall global health measure; patient-reported outcome measure instrument - 29 item survey)
Change in EQ5D3L | preoperatively, postoperatively on day 1 and day 2, week 3 and 6 and 3 months
  relationship between immune markers, actigraphy data using a validated measure of global health state (EQ5D3L)
Change in Edinburgh postnatal depression score (EPDS) | postoperatively on day 2, week 3 and 6 and 3 months
  relationship between immune markers, actigraphy data using a validated measure of depression (EPDS)
Change in Pittsburgh sleep quality index | postoperatively on day 2, week 3 and 6 and 3 months
  relationship between immune markers, actigraphy data using a validated measure of sleep (Pittsburgh sleep index)

CONTACTS AND LOCATIONS:
Overall Officials: Pervez Sultan, MBChB, FRCA, MD(Res), Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No